CLINICAL TRIAL: NCT06144047
Title: Real World Testing and Cost-effectiveness Analysis of Subcutaneous EEG (REAL-ASE)
Brief Title: Real World Testing and Cost-effectiveness Analysis of Subcutaneous EEG
Acronym: REAL-ASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS: 324630
Record Dates: First submitted 2023-11-01; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
Keywords: epilepsy; EEG; subcutaneous EEG; mobile devices; wearable devices
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy (Other): 33 participants with drug-resistant epilepsy will be implanted with the EEGTM SubQ device under local anaesthesia, and will collect 2-channel EEG data, as well as completing an electronic seizure diary, for 6 months
  Interventions: Device: EEG SubQ subcutaneous EEG device

INTERVENTIONS:
Device: EEG SubQ subcutaneous EEG device — 2-channel subcutaneous EEG device

SUMMARY:
The study will investigate whether a novel method to accurately count epileptic seizures, using a CE-marked minimally-invasive ultra long-term subcutaneous electroencephalography (EEG) solution (UNEEG™ SubQ , including 24/7 EEG SubQ), (i) is more accurate than a participant-reported seizure diary; (ii) is feasible and acceptable to participants and clinicians; (iii) reduces impacts of epilepsy and improves quality-of-life; and (iv) provides gains to the healthcare system when rolled-out into the National Health Service (NHS). 33 participants with drug-resistant epilepsy will be implanted with the UNEEG™ SubQ device and will collect data for six months. Annotated seizures from the EEG data will be sent weekly to the treating clinicians, who will communicate with the participants on a monthly basis, and will be free to make any management changes.

ELIGIBILITY:
Key Inclusion Criteria:

* Have given written informed consent
* Diagnosis of treatment-resistant epilepsy of any syndrome in which seizures are detectable in scalp EEG with two electrodes.
* Adults (≥18 years of age)
* Participant routinely keeps a seizure diary, has a smartphone and is willing to use the electronic diary for the study.
* Experiencing ≥10 seizures per year according to their existing seizure diary.
* Willing and able to comply with study procedures

Key Exclusion Criteria:

* Established current diagnosis of psychogenic non-epileptic attacks (dissociative seizures)
* Frequent vigorous involuntary movements (eg. chorea, athetosis) or frequent parasomnias with major motor components (eg. sleep walking, night terrors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of rapid data review of 24/7 EEG SubQ solution | 6 months
  Within-participant correlation between seizure counts per month estimated from rapid review of annotated 24/7 EEG™ SubQ data and 'ground truth' EEG seizure occurrences per month
Diagnostic accuracy of 24/7 EEG SubQ solution compared to diary | 6 months
  Within-participant correlation between seizure counts per month from participant-reported seizure diary and 'ground truth' EEG seizure occurrences per month
Clinician rating of accuracy of 24/7 EEG SubQ | 6 months
  Clinician rating of accuracy of 24/7 EEG SubQ solution

SECONDARY OUTCOMES:
Clinical relevance of the 24/7 EEG SubQ solution | baseline, 2 months and 6 months
  Change over time for average Health Care Professional (HCP) questionnaires 'Communication', 'Insight' & 'Potential of 24/7 EEG™' scores
Proportion of treating clinicians changing clinical management | months 1, 2, 3, 4, 5, 6
  Proportion of treating clinicians changing clinical management throughout the study due to information from the 24/7 EEG SubQ Solution
Participants' perception of the value of receiving feedback about seizure occurrences estimated from EEG data recorded with 24/7 EEG™ SubQ | 6 months
  Participants overall rating of the value of receiving feedback about seizures occurrences every month, across the full study period, from the EEG data recorded with 24/7 EEG™ SubQ
participants' acceptability of real-world implementation with 24/7 EEG™ SubQ Solution | baseline, 2 months and 6 months
  Post-market surveillance questionnaire
Participant adherence with 24/7 EEG™ SubQ Solution | 6 months
  Wear time
Device deficiency | 6 months
  Number of Device deficiencies
EQ-5D-5L score | baseline, 2 months and 6 months
  Change over time for average EQ-5D-5L scores at baseline, 2- months and 6 months
Participant Weighted Quality of Life In Epilepsy (QOLIE-31-P) score | baseline, 2 months and 6 months
  Change over time for average Participant Weighted Quality of Life In Epilepsy (QOLIE-31-P) scores at baseline, 2-months and 6 months
Impact of epilepsy score | baseline, 2 months and 6 months
  Change over time for average Impact of epilepsy score at baseline, 2-months and 6 months
Perceived Self-Mastery Over Epilepsy score | baseline, 2 months and 6 months
  Change over time for average Perceived Self-Mastery Over Epilepsy score at baseline, 2-months and 6 months
health economic impact of epilepsy for participants that have used the 24/7 EEG™ SubQ Solution | 6 months
  Client Services Receipt Inventory (CSRI) scores at 6 months
health economic impact of epilepsy for participants compared to historical controls | 6 months
  Client Services Receipt Inventory (CSRI) score at 6 months compared with the 138 participants in SMILE study in the treatment-as-usual arm
Cost-effectiveness of current practice and 24/7 EEG™ SubQ Solution | 6 months
  Quality-adjusted life-years (QALYs) score
EQ-5D-5L score comparison with historical controls | 6 months
  EQ-5D-5L score compared with the 138 participants in SMILE study in the treatment-as-usual arm
Participant Weighted Quality of Life In Epilepsy (QOLIE-31-P) score comparison with historical controls | 6 months
  Participant Weighted Quality of Life In Epilepsy (QOLIE-31-P) score compared with the 138 participants in SMILE study in the treatment-as-usual arm
Impact of epilepsy score comparison with historical controls | 6 months
  Impact of epilepsy score compared with the 138 participants in SMILE study in the treatment-as-usual arm
Perceived Self-Mastery Over Epilepsy score comparison with historical controls | 6 months
  Perceived Self-Mastery Over Epilepsy score compared with the 138 participants in SMILE study in the treatment-as-usual arm

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Richardson, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided